CLINICAL TRIAL: NCT06323031
Title: Spontaneous Eye Blinking as a Diagnostic and Prognostic Marker in Patients With Disorders of Consciousness After Severe Acquired Brain Injury
Brief Title: Spontaneous Eye Blinking in Disorders of Consciousness
Acronym: Blink-DoC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Therapiezentrum Burgau (Other); University of Liege (Other); University Hospital Munich (Other); Ludwig-Maximilians - University of Munich (Other); VITHAS Valencia (Spain) (Unknown); Lavezzi Susanna, Local Health Unit, Ferrara (IT) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Blink-DoC
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Disorders of Consciousness
Keywords: Disorders of Consciousness; blinking; diagnosis; prognosis; rehabilitation
MeSH Terms: conditions — Consciousness Disorders; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with DoC consecutively admitted to participating units and met the inclusion criteria: Patients in VS or MCS due to severe acquired brain injury with different etiology (traumatic, anoxic, vascular) consecutively admitted at participating neurorehabilitation units. The total sample will be composed of 70 patients (n=9 pts per participating unit).

SUMMARY:
Differential diagnosis between Unresponsive Wakefulness Syndrome (UWS) and Minimally Conscious State (MCS) is complicated due to severe cognitive and/or sensorimotor deficits in these patients. In this study the investigators aimed at exploring the diagnostic and prognostic validity of spontaneous eye blinking parameters (rate, amplitude, duration, variability) in a sample of patients with Disorders of Consciousness (DoC).

This is a multi-center prospective observational study conducted in patients with Severe Acquired Brain Injury (sABI) and DoC admitted to 8 European participating centers, with clinical data collection not deviating from routine practice. The study is non-commercial and will have a maximum total duration of 24 months.

DETAILED DESCRIPTION:
Observational, multicenter, longitudinal study. In this study, all patients admitted to the nine participating centers with diagnosis of DoC, and meeting the inclusion/exclusion criteria, will be enrolled.

The admission of a patient to the research program is subject to the signing of an informed consent by the legal representative/primary caregiver of the patient. The representative will be informed about the study and its objectives, and an informational sheet will be provided.

Population All patients with DoC after sABI consecutively admitted to participating centers who meet the inclusion/exclusion criteria (see below).

Sample size On the basis of the effect size found in a previous study regarding the diagnostic value of eye blink rate (d=0.68), it is planned to enroll 58 patients with DoC (power=0.8; α=0.05) + an additional 20% to cope with possible drop-outs, for a total of 70 patients (23 in UWS, 23 in MCS minus; 23 in MCS plus; about 9 patients per center). For the secondary outcomes (i.e., diagnostic and prognostic value of further blink features) there is no previous data in the literature. In addition, a sample of 23 healthy individuals, balanced in terms of sex and age with the patient sample, will be enrolled as a reference group.

Data collection procedure Within two weeks from study entry, patients will undergo two 20-minute resting electroencephalogram-electrooculogram (EEG-EOG) examinations, separated by 24 hours. Sessions will take place, following standard nursing procedures, between 10:00 AM and 5:00 PM, a time window minimally influenced by circadian peaks of drowsiness in patients with DoC, and a period during which it is believed that EBR is stable in healthy individuals.

The EEG-EOG recording will be conducted at the patient's bedside or, if possible, on their wheelchair, with the patient awake (i.e., eyes open), maintaining a quiet and dimly lit environment. If the patient's arousal level is insufficient, the Coma Recovery Scale-Revised (CRS-R) arousal facilitation protocol will be administered; if the patient continues to keep their eyes closed, the recording session will be postponed to the next available day. During each session, the experimenter is positioned beside the patient, out of her/his visual field. Blinks will be detected in the EOG and defined as a sharp positive peak followed by a negative deflection within a time window of less than 400 ms. To assess the level of consciousness at the time of the EEG-EOG recordings, a CRS-R will be administered at the end of each session. To prevent the patient's awareness of the blink recording from affecting their blink rate, the patient is not informed about the blink recording during the EEG-EOG session but is simply encouraged to remain relaxed with eyes open and not to move. This procedure is carried out independently of the patient's clinical diagnosis. A follow-up assessment is planned at 6 months from T0 (T1).

The healthy volunteers will also perform two resting EEG-EOG examinations, each lasting 20 min, 24 h apart.

EEG will be recorded by at least 19 electrodes placed on the patients' scalp according to the international 10-20 system (Fp1, Fp2, F7, F8, F3, F4, C3, C4, T3, T4, P3, P4, T5, T6, O1, O2, Fz, Cz, Pz) + vertical EOG electrodes, referenced to the vertex. Impedance will be kept below 5 kΩ for electrodes covering the cortex as well as for EOG electrodes. Data will be sampled at a 1000-Hz rate and band pass filtered between 0.1 Hz and 30 Hz; a notch filter will be used to eliminate frequencies around 50 Hz for online visualization. If the EEG recording in a session presents a considerable number of artefacts, the acquisition will be repeated within the next available day.

Enrollment duration: 12 months Study duration: about 24 months.

Statistical plan Patient characteristics at study entry will be compared between the diagnostic groups (UWS, MCS minus, MCS plus) through parametric or non-parametric univariate analyses, as deemed appropriate after verification of data distribution. Similarly, univariate analyses will be performed to compare eye blink rate (EBR) and additional blink features between diagnostic groups.

Univariate within-subject analyses will be performed to compare EBR and additional blink features across time.

In addition, correlation analyses will be performed to verify the existence of a relationship between blink features and level of consciousness as measured by the total score of the CRS-R. If so, logistic regression models will be implemented with blink features and demographic and anamnestic variables as predictors, and outcome as dependent variable. The results will be considered statistically significant if p<05.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of DoC (UWS, MCS minus, MCS plus) following repeated clinical evaluation (at least four CRS-R in a week)
* age ≥ 18 years
* time post-onset ≤6 months
* Previous sABI of any etiology (traumatic, vascular, anoxic, mixed, etc.)
* Negative anamnesis for neurological or psychiatric disorders.

Exclusion Criteria:

* unstable clinical conditions (e.g. respiratory failure, fever, status epilepticus, etc.);
* ophthalmic diseases, or clinically detected peripheral damage in eyelid motility (e.g. orbital fracture);
* intake of sedative drugs in the preceding 24 hours;
* additional brain event following admission (e.g., stroke).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in UWS or MCS due to severe acquired brain injury with different etiology (traumatic, anoxic, vascular) consecutively admitted at participating neurorehabilitation units. The total sample will be composed of 70 patients (n=9 pts per participating unit).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Diagnosis | 6 months from enrollment
  Clinical diagnosis as assessed by the Coma Recovery Scale-Revised (min. - max- score = 0-23, with higher scores indicating a higher level of consciousness)

CONTACTS AND LOCATIONS:
Locations (8):
- Coma Science Group, GIGA-Consciousness, University of Liege, Liège, Belgium, Belgium
- Germany (2):
  - Therapiezentrum Burgau, Burgau, Germany
  - Dipartimento di Neurologia, LMU Hospital, LMU Munich, Munich, Germany
- Italy (4):
  - Polo Specialistico Riabilitativo Fondazione Don Carlo Gnocchi ONLUS, Sant'Angelo dei Lombardi, AV
  - Unità Gravi Cerebrolesioni - Dipartimento Neuroscienze - Azienda Ospedaliera - Universitaria Ferrara, Ferrara, Italy
  - IRCCS Fondazione Don Gnocchi ONLUS, Florence, Italy
  - IRCCS Santa Maria Nascente Fondazione Don Gnocchi ONLUS, Milan, Italy
- Instituto de Rehabilitación Neurológica IRENEA, Valencia, Spain, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request.
Supporting Information: Study Protocol
Time Frame: After study completion.
Access Criteria: Upon reasonable request to the study's PI.

REFERENCES:
- [Background] Wislowska M, Del Giudice R, Lechinger J, Wielek T, Heib DPJ, Pitiot A, Pichler G, Michitsch G, Donis J, Schabus M. Night and day variations of sleep in patients with disorders of consciousness. Sci Rep. 2017 Mar 21;7(1):266. doi: 10.1038/s41598-017-00323-4. PMID 28325926
- [Background] Barbato G, Ficca G, Muscettola G, Fichele M, Beatrice M, Rinaldi F. Diurnal variation in spontaneous eye-blink rate. Psychiatry Res. 2000 Mar 6;93(2):145-51. doi: 10.1016/s0165-1781(00)00108-6. PMID 10725531
- [Background] Magliacano A, Rosenfelder M, Hieber N, Bender A, Estraneo A, Trojano L. Spontaneous eye blinking as a diagnostic marker in prolonged disorders of consciousness. Sci Rep. 2021 Nov 17;11(1):22393. doi: 10.1038/s41598-021-01858-3. PMID 34789832